CLINICAL TRIAL: NCT02366663
Title: SPINOZA / שפינוזה. Study With Preparatory INduction Of Zevalin in Aggressive Lymphoma. A Randomized Phase 3 Study of BEAM Versus 90Yttrium Ibritumomab Tiuxetan (Zevalin) / BEAM in Patients Requiring ASCT for Relapsed DLBCL
Brief Title: BEAM vs. 90-Yttrium Ibritumomab Tiuxetan (Zevalin®)/BEAM With ASCT for Relapsed DLBCL
Acronym: SPINOZA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawal of sponsor support
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12338; NCI-2015-00185 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Non-Hodgkin's lymphoma; autologous stem cell transplantation; radioimmunotherapy; Zevalin; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoma, B-Cell; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type; Antibodies, Monoclonal; Immunologic Factors; Pharmacologic Actions; Physiological Effects of Drugs
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoma, B-Cell; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type | interventions — ibritumomab tiuxetan; Carmustine; Etoposide; Cytarabine; Melphalan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (ZBEAM) (Experimental): Patients receive rituximab IV on days -21 and -14, and 90-yttrium ibritumomab tiuxetan IV on day -14. Patients also receive BEAM comprising carmustine IV over 4 hours on day -6; cytarabine IV over 2 hours BID on days -5 to -2; etoposide IV over 1 hour BID or QD on days -5 to -2; and melphalan IV on day -1. Patients then undergo autologous hematopoietic stem cell transplant on day 0.
  Interventions: Radiation: 90-Yttrium Ibritumomab tiuxetan; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Autologous Hematopoietic Stem Cell Transplant; Biological: Rituximab
- Arm II (BEAM) (Active Comparator): Patients receive BEAM comprising carmustine IV over 4 hours on day -6; cytarabine IV over 2 hours BID on days -5 to -2; etoposide IV over 1 hour BID or QD on days -5 to -2; and melphalan IV on day -1. Patients then undergo autologous hematopoietic stem cell transplant on day 0.
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Autologous Hematopoietic Stem Cell Transplant

INTERVENTIONS:
Radiation: 90-Yttrium Ibritumomab tiuxetan — 0.4 mCi/kg given IV
  Other Names: IDEC Y2B8; Zevalin
  Arms: Arm I (ZBEAM)
Drug: Carmustine — Given IV
  Other Names: BiCNU; FDA 0345
Drug: Etoposide — Given IV
  Other Names: VP-16; Lastet
Drug: Cytarabine — Given IV
  Other Names: Cytosar-U; CHX-3311; U-19920
Drug: Melphalan — Given IV
  Other Names: Alkeran
Procedure: Autologous Hematopoietic Stem Cell Transplant — Autologous Hematopoietic Stem Cell Transplantation (ASCT)
  Other Names: Autologous Stem Cell Transplant
Biological: Rituximab — Given IV
  Other Names: MOAB IDEC-C2B8
  Arms: Arm I (ZBEAM)

SUMMARY:
This randomized phase III trial studies 90-yttrium ibritumomab tiuxetan and combination chemotherapy compared with combination chemotherapy alone before stem cell transplant in treating patients with diffuse large b-cell non-Hodgkin lymphoma that has returned after a period of improvement. Radioactive substances linked to monoclonal antibodies, such as 90-yttrium ibritumomab tiuxetan, can bind to cancer cells and give off radiation which may help kill cancer cells. Drugs used in chemotherapy, such as carmustine, etoposide phosphate, cytarabine, and melphalan (BEAM), work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether 90-yttrium ibritumomab tiuxetan and BEAM before a stem cell transplant are more effective than BEAM alone in treating patients with diffuse large b-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To compare overall survival (OS) between the two transplant arms, with at least a two year of follow-up. SECONDARY OBJECTIVES: I. To compare progression-free survival (PFS), complete response (CR) and partial response (PR) proportion at day 100, time to hematopoietic recovery, incidence of infection, grade III-IV toxicities, treatment-related mortality, incidence of myelodysplastic syndrome (MDS), and secondary acute myelogenous leukemia (AML).

OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive rituximab intravenously (IV) on days -21 and -14, and 90-yttrium ibritumomab tiuxetan IV on day -14. Patients also receive BEAM comprising carmustine IV over 4 hours on day -6; cytarabine IV over 2 hours twice daily (BID) on days -5 to -2; etoposide IV over 1 hour BID or once daily (QD) on days -5 to -2; and melphalan IV on day -1. Patients then undergo peripheral blood stem cell (PBSC) transplant on day 0. ARM II: Patients receive BEAM as in Arm I and undergo PBSC transplant on day 0.

After completion of study treatment, patients are followed up weekly for 30 days, 100 days, 6 months, 1 year, every 3 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD20 positive diffuse large B-cell lymphoma as confirmed by a pathological biopsy report.
2. Patients who are candidates for autologous stem-cell transplantation due to primary refractory or first relapse of disease.
3. Patients must have chemo-sensitive disease achieving at least partial response (Cheson 2007 criteria) to last chemotherapy.
4. Patients with adequate autologous stem cell collection for transplantation (target >= 2.5 x 10^6 CD34+ cells/kg).
5. Patients must sign written informed consent.
6. Adequate birth control in fertile patients.
7. All prior chemotherapy completed at least three weeks before study treatment.
8. Marrow involvement less than 25% at transplantation, no limitation on blood counts (low platelet count allowed).
9. Negative HIV antibody.

Exclusion Criteria:

1. Chemo-refractory disease as determined by less than partial response (Cheson 2007 Criteria) to last chemotherapy.
2. Two or more relapses after initial response to induction chemotherapy.
3. High-grade transformation from earlier diagnosis of low-grade lymphoma. Patients with "De Novo" Transformed DLBCL, defined as DLBCL only on lymph node biopsy and a discordant marrow with para-trabecular small cells at first diagnosis of lymphoma, are eligible if adherent to all other selection criteria.
4. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit.
5. Creatinine > 2.0 mg/dl.
6. KPS < 70.
7. Uncontrolled infection.
8. Pregnancy or lactation.
9. Abnormal lung diffusion capacity (DLCO < 40% predicted).
10. Severe cardiovascular disease; New York Heart Association (NYHA) Functional Classification ≥2.
11. Active CNS disease involvement.
12. Presence of any other malignancy or history of prior malignancy within 5 years of study entry. Within 5 years, patients treated for Stage I or II cancers are eligible provided they have a life expectancy > 5 years in relation to this prior malignance. The 5-year exclusion rule does not apply to-non melanoma skin tumors and in situ cervical cancer.
13. Pleural effusion or ascites > 1 liter.
14. Known hypersensitivity to rituximab.
15. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate.
16. Prior radioimmunotherapy.
17. Prior autologous or allogeneic HSCT.
18. Active evidence of Hepatitis B or C infection; Hepatitis B surface antigen positive.
19. Patients who have had prior radiation to the lung will be excluded from the study, although mediastinal irradiation will be permitted if minimal lung is in the treatment volume.
20. Patients who have received >500cGy radiation to the kidneys will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Y. Krishnan MD, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 69 [66 to 71] | 48 [48 to 48] | 66 [48 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival estimates will be calculated using the Kaplan-Meier method
Time Frame: Measured from randomization to date of death or last follow up date, whichever occurs first, for up to 5 years post randomization
Population: The study was terminated before the data are mature enough to estimate the survival outcome and conduct the test. Therefore, the overall number of participants analyzed is 0 in both groups.
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression-free Survival
Description: Survival estimates will be calculated using the Kaplan-Meier method
Time Frame: Measured from randomization until death, relapse/progression, receipt of anti-lymphoma therapy, or last follow up whichever comes first, for up to 5 years post randomization
Population: as for outcome 1
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Progression
Description: Time-to-event will be measured from the date of ASCT.
Time Frame: Up to 5 years
Population: The study was terminated before the data are mature enough to estimate the cumulative incidence and conduct the test. Therefore, the overall number of participants analyzed is 0 in both groups.
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients With Complete or Partial Response at Day 30
Description: Definition of disease status is based on the article of Revised Response Criteria for Malignant Lymphoma Response Definitions for Clinical Trials (Cheson et al, 2007). Tests used for evaluation of disease status would be physical examination, laboratory testing, bone marrow testing, bone marrow biopsy and aspirate, PET scan, and CT scans of neck, chest, abdomen and pelvis as indicated.
Time Frame: Day 0 to Day +30 post-HCT
Population: In Arm I (ZBEAM), one patient's disease status at Day 30 is not available. Therefore, the overall number of participants analyzed in Arm I (ZBEAM) is 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

5. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be compared between treatment arms using a log-rank test, and the cumulative incidence curves will be estimated.
Time Frame: Day 0 to Day 100 post-HCT
Population: The study was terminated before the data are mature enough to estimate the cumulative incidence and conduct the test. Therefore, the descriptive analysis was performed. The median time to ANC engraftment and range are reported below.
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 2 | 1
days | 11 [11 to 11] | 10 [10 to 10]

6. Secondary Outcome: Incidence of Infection
Description: Microbiologically documented infections will be reported by site of disease, date of onset, severity, and resolution, if any. The incidence of definite and probable viral, fungal and bacterial infections will be tabulated for each patient. The proportion of patients developing infections will be compared between treatment arms.
Time Frame: Day 0 to Day +100 post-HCT
Population: The study was terminated before the data are mature enough to conduct the test. Therefore, the overall number of participants analyzed is 0 in both groups.
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Non-relapse Mortality (NRM) Defined as Death Occurring in a Patient From Causes Other Than Relapse or Progression
Description: The cumulative incidence of NRM will be estimated using the method described by Gooley et al. Differences between cumulative incidence curves in the presence of a competing risk will be tested using the Gray method.
Time Frame: From randomization until non-disease related death, or last follow-up, whichever comes first, assessed up to 5 years
Population: as for outcome 3
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cumulative Incidence of Secondary Malignancies
Description: Incidence of myelodysplastic syndrome (MDS), and secondary acute Myelogenous leukemia (AML) will be compared between the treatment arms using Gray's test.
Time Frame: Up to 5 years
Population: as for outcome 3
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be compared between treatment arms using a log-rank test, and the cumulative incidence curves will be estimated.
Time Frame: Day 0 to Day 100 post-HCT
Population: The study was terminated before the data are mature enough to estimate the cumulative incidence and conduct the test. Therefore, the descriptive analysis was performed. The median time to platelet engraftment and range are reported below.
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 2 | 1
days | 22.5 [19 to 26] | 26 [26 to 26]

10. Secondary Outcome: Number of Patients With Grade 3-5 Toxicities Graded by the NCI CTCAE Version 4.0
Description: Observed toxicities will be summarized in terms of type and severity. In accordance with the secondary study objectives, descriptive analyses on these data will be performed.
Time Frame: Day -21 to Day +100 post-HCT
Population: Number of patients with grade 3, 4 or 5 toxicities in each arm, are reported below.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 2 | 1
Participants
  Anemia | 2 | 1
  Febrile neutropenia | 2 | 1
  Hyperglycemia | 1 | 0
  Hyponatremia | 1 | 0
  INR increased | 1 | 0
  Lymphocyte count decreased | 2 | 1
  Mucositis oral | 2 | 1
  Neutrophil count decreased | 2 | 1
  Obesity | 1 | 1
  Oral pain | 0 | 1
  Pharyngeal mucositis | 0 | 1
  Platelet count decreased | 2 | 1
  Sore Throat | 0 | 1
  White blood cell decreased | 2 | 1

11. Secondary Outcome: Cumulative Incidence of New, Abnormal Cytogenetics
Description: The cumulative incidence of therapy related new, abnormal cytogenetics will be estimated for both groups taking into account the competing risk of death among patients who do not develop a second malignancy.
Time Frame: Day 0 to Year 5 post-HCT
Population: as for outcome 3
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day -21 to Day +100
Description: All the patients who received treatment were assessed periodically for the development of any toxicity. The toxicity rule for safety were assessed as each patient reach Day +30 post-HCT and Day +100 post-HCT. The study PIs, Statisticians and Coordinators reviewed all the Serious Adverse Event occurring in both groups of the trial on an ongoing basis.
Arm/Group | Arm I (ZBEAM) | Arm II (BEAM)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (ZBEAM) (N=2) | Arm II (BEAM) (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Excessive salivation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (2)
Fever (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Mild night sweats (General disorders) | 1 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (3)
Platelet count decreased (Investigations) | 2 (4) | 1 (1)
Weight loss (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 2 (4) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Jitteriness (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (4) | 1 (1)
Hallucinaions (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 2 (4) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Double Vision (Eye disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (4) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
feeling off balance (Nervous system disorders) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
INR increased (Investigations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No